CLINICAL TRIAL: NCT01244035
Title: Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacodynamics and Pharmacokinetics Following Different Dosing Regimens of MK-8266 or Placebo in Subjects With Hypertension
Brief Title: Safety, Pharmacodynamics, and Pharmacokinetics of Different Dosing Regimens of MK-8266 in Participants With Hypertension (MK-8266-008)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 8266-008; 2010-021832-32 (EudraCT Number)
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Results first posted 2019-02-28 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2018-10

CONDITIONS: Hypertension
Keywords: High blood pressure
MeSH Terms: conditions — Hypertension | interventions — BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (12):
- Part I - Sequence ABC (Experimental): Treatment A in Period 1, Treatment B in Period 2, and Treatment C in Period 3
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Part I - Sequence ACB (Experimental): Treatment A in Period 1, Treatment C in Period 2, and Treatment B in Period 3
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Part I - Sequence BCA (Experimental): Treatment B in Period 1, Treatment C in Period 2, and Treatment A in Period 3
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Part I - Sequence BAC (Experimental): Treatment B in Period 1, Treatment A in Period 2, and Treatment C in Period 3
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Part I - Sequence CAB (Experimental): Treatment C in Period 1, Treatment A in Period 2, and Treatment B in Period 3
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Part I - Sequence CBA (Experimental): Treatment C in Period 1, Treatment B in Period 2, and Treatment A in Period 3
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Part II - Sequence DEF (Experimental): Treatment D in Period 1, Treatment E in Period 2, and Treatment F in Period 3
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Part II - Sequence DFE (Experimental): Treatment D in Period 1, Treatment F in Period 2, and Treatment E in Period 3
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Part II - Sequence EFD (Experimental): Treatment E in Period 1, Treatment F in Period 2, and Treatment D in Period 3
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Part II - Sequence EDF (Experimental): Treatment E in Period 1, Treatment D in Period 2, and Treatment F in Period 3
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Part II - Sequence FDE (Experimental): Treatment F in Period 1, Treatment D in Period 2, and Treatment E in Period 3
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F
- Part II -Sequence FED (Experimental): Treatment F in Period 1, Treatment E in Period 2, and Treatment D in Period 3
  Interventions: Drug: Treatment D; Drug: Treatment E; Drug: Treatment F

INTERVENTIONS:
Drug: Treatment A — MK-8266 1.3 mg orally twice daily (BID, 1 mg in the morning and 0.3 mg 8 hours later) plus placebo to match Treatment B on Days 1 through 3. On Day 4, single dose of 1 mg MK-8266.
  Other Names: MK-8266 1.3 mg BID
  Arms: Part I - Sequence ABC; Part I - Sequence ACB; Part I - Sequence BAC; Part I - Sequence BCA; Part I - Sequence CAB; Part I - Sequence CBA
Drug: Treatment B — MK-8266 0.1 mg orally administered every 2 hours as frequent divided dosing (FDD, total dose of 0.9 mg) plus placebo to match Treatment A on Days 1 through 3. On Day 4, single dose of 1 mg MK-8266.
  Other Names: MK-8266 0.9 mg FDD
  Arms: Part I - Sequence ABC; Part I - Sequence ACB; Part I - Sequence BAC; Part I - Sequence BCA; Part I - Sequence CAB; Part I - Sequence CBA
Drug: Treatment C — Placebo to match MK-8266 Treatments A and B orally daily on Days 1 through 3. On Day 4, single dose of placebo to match MK-8266.
  Other Names: Placebo
  Arms: Part I - Sequence ABC; Part I - Sequence ACB; Part I - Sequence BAC; Part I - Sequence BCA; Part I - Sequence CAB; Part I - Sequence CBA
Drug: Treatment D — MK-8266 orally twice daily (1 mg in the morning and 0.4 mg 8 hours later) plus placebo to match Treatment E on Days 1 through 3. On Day 4, single dose of 1 mg MK-8266.
  Arms: Part II - Sequence DEF; Part II - Sequence DFE; Part II - Sequence EDF; Part II - Sequence EFD; Part II - Sequence FDE; Part II -Sequence FED
Drug: Treatment E — MK-8266 0.2 mg orally every 2 hours (total dose of 1.4 mg) plus placebo to match Treatment D on Days 1 through 3. On Day 4, single dose of 1 mg MK-8266.
  Arms: Part II - Sequence DEF; Part II - Sequence DFE; Part II - Sequence EDF; Part II - Sequence EFD; Part II - Sequence FDE; Part II -Sequence FED
Drug: Treatment F — Placebo to match MK-8266 Treatments D and E orally daily on Days 1 through 3. On Day 4, single dose of placebo to match MK-8266.
  Arms: Part II - Sequence DEF; Part II - Sequence DFE; Part II - Sequence EDF; Part II - Sequence EFD; Part II - Sequence FDE; Part II -Sequence FED

SUMMARY:
This was designed as a two part study comprising sequential double-dummy, placebo controlled 3-period randomized crossover studies. The study will evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of different doses and dose regimens of MK-8266. Only Part I of the study was completed.

ELIGIBILITY:
Inclusion Criteria:

* Participant has essential hypertension who is in grade 1 or 2 hypertension according to the European Society of Hypertension (ESH) as delineated in the European Society of Cardiology (ESC) 2007 guidelines, i.e. systolic blood pressure values of 140-179 and diastolic blood pressure values of 90-109 on at least 3 occasions prior to the study.
* Otherwise healthy participants with grade 1 or 2 arterial hypertension who are treated with a single antihypertensive drug and meet the above blood pressure criteria may be enrolled at the discretion of the investigator
* Participant is generally in good health with the exception of hypertension
* Participant is a nonsmoker and/or has not used nicotine or nicotine-containing products for 6 months

Exclusion Criteria:

* Participant has a history of any illness that might confound the results of the study or pose and additional risk to the participant if they take part in the study
* Participant has a history of stroke, chronic seizures, or major neurological disorder
* Participant has a disability that can interfere with rising from a semi-recumbent position to the standing position
* Participant has a personal or family history of a bleeding or clotting disorder
* Participant has a history of frequent nosebleeds or recurrent or active gingivitis
* Participant has a history of cancer, except 1) certain skin cancers; 2) cancer successfully treated more than 10 years prior to the study that has not recurred; or, 3) participants who are unlikely to have a recurrence during the study
* Participant has a history of cardiac disease including but not limited to heart valve disease or evidence of secondary cardiac damage
* Participant is categorized as class II or greater according to the New York Heart Association (NYHA) functional classification for heart failure
* Participant is unable to refrain from use of prescription or non-prescription drugs or herbal remedies (such as St. John's Wort) during the study
* Participant anticipates using phosphodiesterase (PDE5) inhibitors [sildenafil (Viagra®), tadalafil (Cialis®), or vardenafil (Levitra®)] during the study
* Participant consumes excessive amounts of alcohol (more than 3 drinks per day) or caffeine (more than 6 servings a day)
* Participant has had major surgery, donated or lost 1 unit of blood, or participated in another investigational within 4 weeks prior to the study
* Participant has a history of multiple and/or severe allergies, or has had an anaphylactic reaction or intolerance to any drugs or food

Ages: 21 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2010-08-19 (Actual); Primary Completion 2010-12-23 (Actual); Study Completion 2010-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinicaltrials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The same participants in Part 1 were to continue in Part 2, pending the planned evaluation of Part 1 pharmacodynamic results. Based on the Part 1 results, no participants continued to Part 2.
Groups:
- Sequence ABC: MK-8266 1.3 mg BID, then MK-8266 0.9 mg FDD, then Placebo
- Sequence ACB: MK-8266 1.3 mg BID, then Placebo, then MK-8266 0.9 mg FDD
- Sequence BCA: MK-8266 0.9 mg FDD, then Placebo, then MK-8266 1.3 mg BID
- Sequence BAC: MK-8266 0.9 mg FDD, then MK-8266 1.3 mg BID, then Placebo
- Sequence CAB: Placebo, then MK-8266 1.3 mg BID, then MK-8266 0.9 mg FDD
- Sequence CBA: Placebo, then MK-8266 0.9 mg FDD, then MK-8266 1.3 mg BID
Period: Part 1: Period 1
Arm/Group | Sequence ABC | Sequence ACB | Sequence BCA | Sequence BAC | Sequence CAB | Sequence CBA
Started (This was a 3-period crossover study with a 4-day washout between treatment periods) | 5 | 5 | 6 | 5 | 5 | 5
Completed | 4 | 3 | 4 | 5 | 4 | 3
Not Completed | 1 | 2 | 2 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Fulfilled Stopping Criteria | 1 | 0 | 2 | 0 | 1 | 1
Period: Part 1: Period 2
Arm/Group | Sequence ABC | Sequence ACB | Sequence BCA | Sequence BAC | Sequence CAB | Sequence CBA
Started | 4 | 3 | 4 | 5 | 4 | 3
Completed | 4 | 3 | 3 | 5 | 4 | 3
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Fulfilled Stopping Criteria | 0 | 0 | 1 | 0 | 0 | 0
Period: Part 1: Period 3
Arm/Group | Sequence ABC | Sequence ACB | Sequence BCA | Sequence BAC | Sequence CAB | Sequence CBA
Started | 4 | 3 | 3 | 5 | 4 | 3
Completed | 4 | 2 | 3 | 5 | 3 | 2
Not Completed | 0 | 1 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Deviation | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This was a 3-period crossover study, with a total of 31 randomized participants at Baseline in Sequences A, B, and C.
Groups:
- All Participants, All Sequences: A: MK-8266 1.3 mg BID, B: MK-8266 0.9 mg FDD, C: Placebo
Arm/Group | All Participants, All Sequences
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Total of 31 participants in Sequences A, B, and C
  Years | 49.1 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 31
Heart Rate (HR) [Mean (Standard Deviation); unit: Beats per minute] — HR summary for the enrolled population Population: All participants who were randomized to receive study treatment and had HR measurement
  Beats per minute | 78.00 (8.77)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] — DBP summary for the enrolled population Population: All participants who were randomized to receive study treatment and had DBP measurement
  mmHg | 93.36 (5.08)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events (AEs)
Description: The number of participants with one or more clinical or laboratory AEs was assessed. An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product.
Time Frame: MK-8266 1.3 mg BID and 0.9 mg FDD groups: Up to Day 4 in each period; MK-8266 1 mg QD group: the last AE was reported on day 10 after the last dose; Placebo group: Up to 10-14 days after the last dose of placebo
Population: All participants who received at least one dose of study treatment
Measure: Count of Participants; unit: Participants
Groups:
- MK-8266 1.3 mg BID: Participants receiving MK-8266 1.3 mg BID on Day 1 - Day 3, and MK-8266 1 mg as a single dose on Day 4.
- MK-8266 0.9 mg FDD: Participants receiving MK-8266 0.9 mg BID on Day 1 - Day 3, and MK-8266 1 mg as a single dose on Day 4.
- MK-8266 1 mg QD: Participants receiving MK-8266 administered as a single 1 mg dose on Day 4.
- Placebo: Participants receiving placebo matching MK-8266 administered on Days 1, 2, 3 and 4.
Arm/Group | MK-8266 1.3 mg BID | MK-8266 0.9 mg FDD | MK-8266 1 mg QD | Placebo
Number analyzed (Participants) | 25 | 26 | 26 | 27
Participants | 9 | 16 | 8 | 9

2. Primary Outcome: Area Under the MK-8266 Concentration Versus Time Curve AUC(0-8 Hours) on Days 1 and 3
Description: The AUC(0-8 hours) of MK-8266 was assessed. The arithmetic mean and standard deviation values of AUC(0-8 hours), based on the raw scale, are provided.
Time Frame: Pre-dose and 0.5, 1, 2, 4, and 8 hours after dosing on Day 1, and pre-dose and 4 and 8 hours after dosing on Day 3 of each period
Population: All participants who received at least one dose of the investigational drug and had assessment of AUC(0-8 hours)
Measure: Mean (Standard Deviation); unit: nM*hr
Groups:
- MK-8266 1.3 mg BID; MK-8266 1 mg QD: Participants receiving MK-8266 1.3 mg BID on Day 1 - Day 3, and MK-8266 1 mg as a single dose on Day 4.
- MK-8266 0.9 mg FDD; MK-8266 1 mg QD: Participants receiving MK-8266 0.9 mg FDD on Day 1 - Day 3, and MK-8266 1 mg as a single dose on Day 4.
Arm/Group | MK-8266 1.3 mg BID; MK-8266 1 mg QD | MK-8266 0.9 mg FDD; MK-8266 1 mg QD
Number analyzed (Participants) | 24 | 24
nM*hr
  Day 1 | 83.4 (22.2) | 23.7 (5.96)
  Day 3 | 120 (41.7) | 69.3 (25.8)

3. Primary Outcome: Area Under the MK-8266 Concentration Versus Time Curve AUC(0-8 Hours) on Day 4
Description: as for outcome 2
Time Frame: Predose and 2, 4, and 8 hours after dosing on Day 4 of each period
Population: All participants who received at least one dose of the investigational drug and had assessment of AUC(0-8 hours)
Measure: Mean (Standard Deviation); unit: nM*hr
Arm/Group | MK-8266 1.3 mg BID; MK-8266 1 mg QD | MK-8266 0.9 mg FDD; MK-8266 1 mg QD
Number analyzed (Participants) | 24 | 24
nM*hr | 135 (46.6) | 139 (43.2)

4. Primary Outcome: Maximum Plasma Concentration (Cmax) of MK-8266 on Day 1 and Day 3
Description: The Cmax of MK-8266 was assessed. The arithmetic mean and standard deviation values of Cmax, based on the raw scale, are provided.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8, 12, 14, 15, and 16 hours after dosing on Days 1 and 3
Population: All participants who received at least one dose of the investigational drug and had assessment for Cmax
Measure: Mean (Standard Deviation); unit: mg/mL
Groups:
- MK-8266 1.3 mg BID; MK-8266 0.9 mg FDD: All Treatment Sequences (A, B, C) for Day 1 to Day 3
Arm/Group | MK-8266 1.3 mg BID | MK-8266 0.9 mg FDD
Number analyzed (Participants) | 24 | 24
mg/mL
  Day 1 | 17.4 (4.01) | 8.63 (2.85)
  Day 3 | 20.5 (6.11) | 11.0 (3.73)

5. Primary Outcome: Maximum Plasma Concentration (Cmax) of MK-8266 on Day 4
Description: as for outcome 4
Time Frame: Predose and 2, 4, and 8 hours after dosing on Day 4 of each period
Population: All participants who received at least one dose of the investigational drug and had assessment for Cmax
Measure: Mean (Standard Deviation); unit: nM
Groups:
- MK-8266 0.9 mg FDD; MK-8266 1 mg QD: Participants receiving MK-8266 1.3 mg BID on Day 1 - Day 3, and MK-8266 1 mg as a single dose on Day 4.
Arm/Group | MK-8266 1.3 mg BID; MK-8266 1 mg QD | MK-8266 0.9 mg FDD; MK-8266 1 mg QD
Number analyzed (Participants) | 24 | 24
nM | 23.1 (7.28) | 23.3 (6.86)

6. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of MK-8266 on Day 1 and Day 3
Description: The Tmax of MK-8266 was assessed. Descriptive statistics are provided for the minimum, median and maximum values for the Tmax of MK-8266 on Day 1 and Day 3.
Time Frame: Pre-dose and 0.5, 1, 2, 4, 8, 12, 14, 15, and 16 hours after dosing on Days 1 and 3
Population: All participants who received at least one dose of the investigational drug and had assessment for Tmax
Measure: Median (Full Range); unit: Hours
Arm/Group | MK-8266 1.3 mg BID | MK-8266 0.9 mg FDD
Number analyzed (Participants) | 24 | 24
Hours
  Day 1 | 4.0 [2.0 to 12.0] | 16.0 [8.0 to 24.0]
  Day 3 | 4.0 [4.0 to 12.0] | 16.0 [4.0 to 24.0]

7. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of MK-8266 on Day 4
Description: The Tmax of MK-8266 was assessed. Descriptive statistics are provided for the minimum, median and maximum values for the Tmax of MK-8266 on Day 4.
Time Frame: Predose and 2, 4, and 8 hours after dosing on Day 4 of each period
Population: All participants who received at least one dose of the investigational drug and had assessment for Tmax
Measure: Median (Full Range); unit: Hours
Groups:
- MK-1.3 mg BID; MK-8266 1 mg QD: Participants receiving MK-8266 1.3 mg BID on Day 1 - Day 3, and MK-8266 1 mg as a single dose on Day 4.
- MK-8266 0.9 mg FDD, MK-8266 1 mg QD: Participants receiving MK-8266 0.9 mg FDD on Day 1 - Day 3, and MK-8266 1 mg as a single dose on Day 4.
Arm/Group | MK-1.3 mg BID; MK-8266 1 mg QD | MK-8266 0.9 mg FDD, MK-8266 1 mg QD
Number analyzed (Participants) | 24 | 24
Hours | 4.0 [2.0 to 8.0] | 4.0 [2.0 to 8.0]

8. Primary Outcome: Change From Baseline in Heart Rate (HR)
Description: The effect of MK-8266 and placebo on changes in HR were assessed, as measured by time weighted average change from baseline in HR over 0-24 hours postdose (TWA^0-24 hr) on Day 3. Baseline values for HR are shown in the Baseline Characteristics section.
Time Frame: Pre-dose (Baseline) and every 30 minutes for the first 4 hours, followed by hourly up to 24 hours after dosing on Day 3
Population: All participants who received at least one dose of the investigational drug and had HR measurements
Measure: Least Squares Mean (Standard Deviation); unit: Beats per minute
Groups:
- MK-8266 0.9 mg FDD: MK-8266 administered as 0.1 mg every 2 hours (total dose of 0.9 mg) on Days 1, 2, and 3
- MK-8266 1.3 mg BID: MK-8266 administered as 1.0 mg in the morning + 0.3 mg 8 hours later on Days 1, 2, and 3
- Placebo: Matching placebo administered at time points matching administration of MK-8266 on Days 1, 2, and 3
Arm/Group | MK-8266 0.9 mg FDD | MK-8266 1.3 mg BID | Placebo
Number analyzed (Participants) | 25 | 24 | 25
Beats per minute | 2.78 (6.67) | 5.84 (3.94) | 1.68 (3.67)
Statistical Analysis 1: Comparison: MK-8266 0.9 mg FDD vs Placebo; Test type: Other; p = 0.1325, Linear mixed effects model; Period and treatment were fixed effects and participant was a random effect; LS Mean difference = 1.10, 90% CI 2-sided [-0.54 to 2.74]
Statistical Analysis 2: Comparison: MK-8266 1.3 mg BID vs Placebo; Test type: Other; p < 0.001, Linear mixed effects model; Period and treatment were fixed effects and participant was a random effect; LS Mean difference = 4.16, 90% CI 2-sided [2.53 to 5.79]
Statistical Analysis 3: Comparison: MK-8266 0.9 mg FDD vs MK-8266 1.3 mg BID; Test type: Other; p = 0.0016, Linear mixed effects model; Period and treatment were fixed effects and participant was a random effect; LS Mean difference = -3.06, 90% CI 2-sided [-4.70 to -1.42]

9. Primary Outcome: Change From Baseline in Diastolic Blood Pressure (DBP)
Description: The effect of MK-8266 and placebo on changes in diastolic blood pressure (DBP) were assessed, as measured by time weighted average change from baseline in DBP over 0-24 hours postdose (TWA^0-24 hr) on Day 3. Baseline values for DBP are shown in the Baseline Characteristics section.
Time Frame: Pre-dose (Baseline) and every 30 minutes for the first 4 hours, followed by hourly up to 24 hours after dosing on Day 3
Population: All participants who received at least one dose of the investigational drug and had DBP measurements.
Measure: Least Squares Mean (Standard Deviation); unit: mmHg
Arm/Group | MK-8266 0.9 mg FDD | MK-8266 1.3 mg BID | Placebo
Number analyzed (Participants) | 25 | 24 | 24
mmHg | -3.21 (3.77) | -3.04 (5.30) | -0.28 (4.68)
Statistical Analysis 1: Comparison: MK-8266 0.9 mg FDD vs Placebo; Test type: Other; p = 0.0212, Linear mixed effects model; Period and treatment were fixed effects and participant was a random effect; LS Mean difference = -2.94, 90% CI 2-sided [-5.30 to -0.57]
Statistical Analysis 2: Comparison: MK-8266 1.3 mg BID vs Placebo; Test type: Other; p = 0.0299, Linear mixed effects model; Period and treatment were fixed effects and participant was a random effect; LS Mean difference = -2.76, 90% CI 2-sided [-5.16 to -0.36]
Statistical Analysis 3: Comparison: MK-8266 0.9 mg FDD vs MK-8266 1.3 mg BID; Test type: Other; p = 0.4506, Linear mixed effects model; Period and treatment were fixed effects and participant was a random effect; LS Mean difference = -0.18, 90% CI 2-sided [-2.54 to 2.19]

ADVERSE EVENTS:
Time Frame: MK-8266 1.3 mg BID and 0.9 mg FDD groups: Up to Day 4 in each period; MK-8266 1 mg QD group: the last AE is reported on day 10 after the last dose; Placebo group: Up to 10-14 days after the last dose of placebo
Groups:
- MK-8266 0.9 mg FDD: MK-8266 administered as 0.1 mg every 2 hours on Days 1, 2, and 3
- MK-8266 1 mg QD: MK-8266 administered a single 1 mg dose on Day 4
- Placebo: Placebo matching MK-8266 administered on Days 1, 2, 3 and 4
Arm/Group | MK-8266 1.3 mg BID | MK-8266 0.9 mg FDD | MK-8266 1 mg QD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/26 | 0/26 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26 | 0/26 | 0/27
Other Adverse Events (participants affected / at risk) | 9/25 | 16/26 | 8/26 | 9/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8266 1.3 mg BID (N=25) | MK-8266 0.9 mg FDD (N=26) | MK-8266 1 mg QD (N=26) | Placebo (N=27)
Accelerated idioventricular rhythm (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Open wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (8)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 1 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (3)
Headache (Nervous system disorders) | 4 (6) | 5 (5) | 2 (2) | 3 (4)
Hemicephalalgia (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nervousness (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.